CLINICAL TRIAL: NCT05435053
Title: Irreversible Electroporation in Combination With Immune Checkpoint Inhibition, in Patients With Metastatic Pancreatic Cancer - A Prospective, Phase 2 Study
Brief Title: Irreversible Electroporation + Nivolumab for Patients With Metastatic Pancreatic Cancer
Acronym: CHECKPOINT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on the basis on an evaluation of the safety and efficacy of the 9 included patients of which 2 of the patients were excluded before receiving any study treatments, thus 7 patients were treated in the study.
Sponsor: Ismail Gögenur (Other)
Responsible Party: Sponsor-Investigator, Ismail Gögenur, Professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26092020; 2020-004623-17 (EudraCT Number)
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pancreas Cancer
Keywords: Irreversible electroporation; Immunotherapy; Nivolumab; Abscopal effect
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- IRE + Nivolumab (Experimental): IRE on Day 1, followed by Nivolumab on Day 2/3 and then every 2 weeks (q2w) for a maximum of 24 weeks.
  Interventions: Drug: Nivolumab; Device: Irreversible electroporation (IRE)

INTERVENTIONS:
Drug: Nivolumab — Every 2 weeks (3 mg/kg, maximum of 240 mg) for up to 24 weeks
  Nivolumab is an immune checkpoint inhibitor (PD-1-inhibitor).
  Other Names: Opdivo
Device: Irreversible electroporation (IRE) — Percutaneous ablation of a primary in-situ (or locally-recurrent) or metastatic lesion.
  Irreversible electroporation is delivered through the NanoKnife system (AngioDynamics, New York, USA). The system is FDA-approved for medical use.

SUMMARY:
The trial investigates the safety and efficacy of irreversible electroporation in combination with checkpoint inhibition in patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
The trial is designed as an investigator initiated prospective phase 2 study in patients with metastatic pancreatic cancer (PC) to determine the efficacy and safety of checkpoint inhibition administered concurrently with irreversible electroporation.

A recently published preclinical study by Zhao et al. (2019) showed that the combination of IRE and PD-1-inhibitor suppressed the tumour growth and increased the survival of mice bearing pancreatic cancer.

The aim of the trial is to initiate an abscopal response, leveraging the patient's immune system in eliciting a sufficient immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Histopathological confirmation of pancreatic adenocarcinoma.
3. At least one measurable primary in-situ (or locally-recurrent) or metastatic tumor must be present and, in the opinion of the investigators be amenable to IRE, and at least one additional metastatic tumor that will not undergo IRE. Both lesions must be accessible for image-guided percutaneous biopsy.
4. Age > 18 years
5. Life expectancy greater than 3 months
6. ECOG (Eastern Cooperative Oncology Group) Performance Status (PS) 0-1
7. Patients must have normal organ and marrow function as defined below:

   * White blood cell count (WBC) ≥ 2 x 10⁹/L
   * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
   * Hemoglobin ≥ 5,6 mmol/l
   * Platelet count ≥ 100 x 10⁹/L
   * Serum bilirubin ≤1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L )
   * ASAT/ALAT ≤3 x ULN ( < 5 x ULN if known liver metastasis)
   * PP ≥ 40 or INR ≤ 1.5
   * Serum creatinine ≤ 1.5 x ULN or eGFR ≥ 40 mL/min
8. Women of childbearing potential (WOCBP) must use method(s) of contraception as indicated per protocol.
9. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab.
10. Women must not be breastfeeding
11. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year.
12. Men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug.

Exclusion Criteria:

1. Malignant ascites that is clinically detectable by physical examination or is symptomatic.
2. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or checkpoint pathways
3. Radiotherapy, or major surgery within the last 2 weeks prior to entering the study
4. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
5. Patients should be excluded if they have an active, known or suspected autoimmune disease.
6. Patients should be excluded if they are positive test for hepatitis B virus surface anti-gen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
7. Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immuno-suppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
8. PD-1 inhibitors may cause hepatic toxicity which may lead to caution regarding other potentially hepatotoxic drugs.
9. Allergies and Adverse Drug Reaction

   * History of allergy to study drug components
   * History of severe hypersensitivity reaction to any monoclonal antibody
10. Patients are excluded if they have active brain metastases or leptomeningeal metastases. Subjects with brain metastases are eligible if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for [lowest minimum is 4 weeks or more] after treatment is complete and within 28 days prior to the first dose of nivolumab administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
11. Contraindications for IRE:

    * Implanted pacemaker or ICD (Implantable cardioverter defibrillator) unit.
    * History of epilepsy
    * History of cardiac arrhythmia
    * Recent myocardial infarction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events [Safety and Tolerability] | 6 months after start of treatment
  Determined by the incidence and severity of treatment related adverse events according to CTCAE version 4.0

SECONDARY OUTCOMES:
Tumor response by CT | Baseline compared to 3 and 6 months after start of treatment
  Based on CT chest/abdomen scans according to RECIST version 1.1
Tumor response by ultrasound | Baseline compared to 3 and 6 months after start of treatment
  Based on contrast enhanced ultrasound (CEUS) utilizing the standardized and quantitative method Dynamic CEUS (DCEUS)
Progression free survival | From start of treatment until unequivocal disease progression, assessed up to 5 years
  In terms of months
Overall survival | From start of treatment until unequivocal disease progression, assessed up to 5 years
  In terms of months
Quality of life using EORTC QLQ-C30 | Baseline compared to 14 days, 3 and 6 months after start of treatment
  EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, Professor, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No